CLINICAL TRIAL: NCT02333019
Title: A Parent Child Program to Prevent Adolescent Pregnancy
Acronym: PPP_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Schroeder, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SBIR79RR-IIRR; R44HD048057 (NIH)
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Adolescent Pregnancy; Sexually Transmitted Diseases; Parental; Communication; Sexuality
Keywords: risk
MeSH Terms: conditions — Sexually Transmitted Diseases; Communication; Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Let's Talk About Sex (Experimental): Participants assigned to the treatment condition viewed a multimedia web site designed to help parents of pre-adolescent children, aged 10 to 14 years old, build skills to communicate effectively about parental values and issues relating to sexuality, sex and relationships, and preventing pregnancy and sexually transmitted infections.
  Interventions: Behavioral: Let's Talk About Sex
- Websites; preventing teen pregnancy (Active Comparator): Participants assigned to the control condition were emailed urls for websites with information similar to the Let's Talk about Sex program. Parents were directed to the parents section of the National Campaign to Prevent Teen and Unplanned Pregnancy and children were directed to Nemours' KidsHealth website.
  Interventions: Behavioral: Websites; preventing teen pregnancy

INTERVENTIONS:
Behavioral: Let's Talk About Sex — Multimedia web site to build parental skills in communicating with their pre-adolescnet child sex and relationships, pregnancy prevention, and risk of sexually transmitted infections.
  Arms: Let's Talk About Sex
Behavioral: Websites; preventing teen pregnancy — Two general web sites with information about preventing teen pregnancy
  Arms: Websites; preventing teen pregnancy

SUMMARY:
While the U.S. teen birth rate is currently at its lowest level, it remains high in relation to other industrialized countries and continues to be a public health concern due to health risks for teen mothers and their babies, and associated social and economic costs. Parental monitoring, supervision, and open communication about sexual issues have been found to be protective factors for adolescent sexual activity and pregnancy. Our theoretically based Internet program for parents of pre-adolescent children aged 10-14, Let's Talk about Sex, is designed to build parental communication, knowledge, and attitudes to discuss sensitive topics with their child, including sexuality, pregnancy prevention, and preventing sexually transmitted illnesses (STIs). This age group of children was selected because parental communication about pregnancy and STI prevention will be most effective if initiated prior to, rather than after, the age when children commonly become sexually active. The "Let's Talk about Sex" program is grounded in behavior change theory and incorporates the use of video for behavioral modeling and emotional support.

DETAILED DESCRIPTION:
"Let's Talk about Sex" was designed to help parents talk to their 10- to 14-year old children about sex and relationships. The goal of the program for the parent was to build skills to communicate effectively with their children about parental values and about issues relating to sexuality, specifically by: a) increasing communication with their child about sexuality; b) increasing behavioral intentions to communicate; c) decreasing perceived barriers to communicating about sexuality; (d) increasing perceived sense of importance/motivation for communicating about sexuality; and e) increasing knowledge about risks of adolescent pregnancy and sexually transmitting infections (STIs). The goal of the intervention for the child was to increase child-parent communication about sexuality issues.

Program content was derived from the research literature; focus group findings, and input from professional consultants, experts in the field with extensive experience working with communication about sexuality. Modifications to content and program format were made based on iterative usability testing.

The parents' program was structured around five sessions, which guided the user through a topic-oriented experience of the content. The program used text, video narration, and video testimonials to present the intervention material. Emails were sent to users weekly for 8 weeks, with a link to a recommended session. Users could also browse the content freely as desired. Topics for parents included (1) Influencing your child's decisions about sex; (2) Understanding your own sexual values and beliefs; (3) Helping your child prepare for adolescence; (4) Preventing pregnancy and disease; and (5) Healthy relationships. Parents who responded to a values and beliefs quiz within the "Understanding your own sexual values and beliefs" section were presented with recommended articles tailored to their responses.

The child's intervention was structured as one session with four brief topics: (1) a whiteboard animation titled "How to talk to your parents about sex and not die of embarrassment"; (2) an article about bodily changes related to puberty; (3) a "What's most important to me" quiz; and (4) an article about healthy relationships.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian with a child 10-14 years of age
* Parent / guardian must be over the age of 18
* Child must live with the parent participating in the study at least 50% of the time

Exclusion Criteria:

* Parents or guardians with a child not fitting within the specified age range
* Parents or guardians whose child does not live with him/her at least 50% of the time
* Parents or guardians younger than 18 years old; due to online nature of the evaluation, we were unable to verify parental consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Behavioral activation as measured by the Parent-Teen Sexual Risk Communication Scale | 8-week follow-up
  Behavioral activation around discussions with their child was assessed with 9 items from the Parent-Teen Sexual Risk Communication Scale (Hutchinson, 2007). The items measure the type and quantity of information relayed in the parent-child conversation and were adapted to more precisely measure the content of the program (e.g., In general how much information have you shared with your daughter or son about human sexuality?). Response options were on a 5-point scale (1=none; 5=everything).

SECONDARY OUTCOMES:
Behavioral intentions of parent to communicate with their child about sexuality and related topics | 4-week posttest and 8-week follow-up
  Seven items measuring parental intentions to talk with their child about sexuality, relationships, dating, preventing pregnancy and STSIs were derived from the content of the program (e.g., How likely is it that you will talk to your child about your values and beliefs about sex and relationships?). Response options were on a 5-point scale (1=extremely unlikely; 5=extremely likely).
Parents' perceived barriers in communicating with their children regarding pregnancy prevention and contraception | 4-week posttest and 8-week follow-up
  Attitudes and beliefs around barriers were assessed with a 16- item scale developed by Jaccard et al. (2000) to measure beliefs, attitudes, and perceived barriers to parents communicating with children regarding pregnancy prevention and contraception. Items were adapted to more precisely measure the content of the program (e.g., My child is just too busy to talk to me about sex and birth control). Response options were on a 5-point scale (1=strongly disagree; 5=strongly agree).
Parents' perception of importance of communicating with their teen about sexuality and related topics | 4-week posttest and 8-week follow-up
  Attitudes and beliefs around importance/motivation were assessed with a 6-item scale developed from concepts taught in the program pertaining to parents' sense of importance or motivation for communicating with their teen about sexuality (e.g., It is extremely important to me to talk to my child about his/her sexual feelings.). Response options were on a 5-point scale (1=strongly disagree; 5=strongly agree).
Parents' knowledge of parent-teen communication about sexuality, birth control, and preventing sexually transmitted infections. | 4-week posttest and 8-week follow-up
  A 10-item true-false scale and 5 multiple-choice items were developed from program content to assess parents' knowledge of parent-teen communication about sexuality, birth control, and preventing STIs. The total number of correct items was divided by the total number of items representing the proportion of knowledge items correctly endorsed.
Users' perception of program usability | 4-week posttest
  At posttest (T2), treatment participants completed an 11-item questionnaire from the Action-WAMMI (Chambers et al., 2002) assessing ease of use and experience in the program. Users were asked to what degree they agreed or disagreed with program use and satisfaction statements on a 5-point scale (1=strongly disagree; 5=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Schroeder, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States